CLINICAL TRIAL: NCT01326741
Title: Detection of Clonal Mast Cell Disorders Among Patients With Exercise-induced Anaphylaxis
Brief Title: Clonal Mast Cell Disorders in Exercise-Induced Anaphylaxis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Cem Akin, MD, PhD, Brigham and Women's Hospital
Other Study IDs: 2010P002042
Record Dates: First submitted 2011-03-29; First posted 2011-03-31 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Anaphylaxis
Keywords: clonal mast cell disorder; exercise-induced anaphylaxis; hypotension
MeSH Terms: conditions — Anaphylaxis; Exercise-Induced Allergies; Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Anaphylaxis is a serious allergic reaction that develops rapidly and can cause death. Some patients experience anaphylaxis is association with exercise, a disorder called exercise-induced anaphylaxis. A subset of patients with unexplained anaphylaxis, especially those with hypotension during the anaphylactic episodes, have been shown to have abnormal, clonal populations of a certain cell type, mast cells, in the bone marrow. This has been described in at least one patient with exercise-induced anaphylaxis. The investigators would like review the findings in a group of patients with exercise-induced anaphylaxis who have undergone evaluation for the presence of abnormal, clonal mast cells.

ELIGIBILITY:
Inclusion Criteria:

* Anaphylaxis in association with exercise on at least two occasions
* During anaphylactic reaction, the subject must have experienced one or more of the following: flushing, hypotension, lack of urticaria

Exclusion Criteria:

* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ten adults of either sex
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2011-03

PRIMARY OUTCOMES:
Number of participants with presence of clonal abnormalities in the bone marrow specimen | Baseline
  Presence of clonal mast cells in bone marrow as assessed by D816V c-kit mutation or CD25 will be recorded for each participant.
Number of participants with presence of clonal abnormalities in the bone marrow specimen | Baseline
  Presence of clonal mast cells in bone marrow as assessed by D816V c-kit mutation or CD25 will be recorded for each participant. The data will be reported as the number of participant with exercise induced anaphylaxis carrying these clonal mast cells in this observational study. Presence of mast cells will be correlated with clinical parameters such as symptoms experienced during anapylaxis.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Akin C, Scott LM, Kocabas CN, Kushnir-Sukhov N, Brittain E, Noel P, Metcalfe DD. Demonstration of an aberrant mast-cell population with clonal markers in a subset of patients with "idiopathic" anaphylaxis. Blood. 2007 Oct 1;110(7):2331-3. doi: 10.1182/blood-2006-06-028100. Epub 2007 Jul 16. PMID 17638853